CLINICAL TRIAL: NCT06342492
Title: Conduction System Vs Surgical Left Ventricular Epicardial Pacing For Coronary Sinus Lead Failure
Status: Recruiting | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRRF_CS Lead Failure_0025
Record Dates: First submitted 2024-02-06; First posted 2024-04-02 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conduction System Pacing: Subjects who had lead placement via conduction system pacing approach
  Interventions: Other: Coronary Sinus Lead Revision
- Epicardial Lead Placement: Subjects who had lead placement via transthoracic, epicardial approach
  Interventions: Other: Coronary Sinus Lead Revision

INTERVENTIONS:
Other: Coronary Sinus Lead Revision — Coronary Sinus Lead Revision

SUMMARY:
This a single-center, retrospective, observational study of patients that undergo coronary sinus(CS) lead revision, comparing epicardial lead placement to coronary sinus pacing(CSP) in those that had lead failure.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy with defibrillator(CRT-D) improves quality of life, functionality, and even mortality for select patients with severe heart failure with reduced ejection fraction (HFrEF). It traditionally consists of three leads placed endovascularly into the right atrium, right ventricle, and left ventricle (LV) [typically placed into the CS], known as biventricular pacing resynchronization (BVP-CRT), respectively, from which electrical stimulation enables improved cardiac synchrony. Nonetheless, the placement of a CRT-D is not without risks. Lead-related complication is high and CRT-D implantation fails in up to 30% of patients due to lead placement alone.

Epicardial lead placement and CSP have been deemed viable alternatives to CRT-D. It has even been shown to be options in patients that fail conventional BVP-CRT. This is primarily due to increased accuracy, decreased complications, and even durability. However, guidelines for decision between a transthoracic approach and CSP is unclear, even more so after lead failure. Instead, this decision is currently individualized to the patient. There is a lack of prospective and head-to-head data between the two, and this study is aimed to compare transthoracic LV epicardial lead placement and CSP in patients with lead failure after BVP-CRT.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years of age
* Patients with HFrEF that underwent BVP-CRT
* Experienced CS lead failure, whether initial or recurrent, subsequently replaced with transthoracic epicardial lead placement or CSP
* Underwent Medtronic, Boston Scientific, or Abbott lead placement

Exclusion Criteria:

* Patients younger than 18 years of age
* Transthoracic epicardial lead placement or CSP performed as the initial approach or for other reasons than lead replacement
* Those for which CRT no longer provides symptom relief or mortality benefit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who underwent CS lead revision, comparing epicardial lead placement to CSP in those that had lead failure.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Need for lead revision | Procedure Day
  Compare the need for lead revision between conduction system pacing (CSP) and transthoracic left ventricular (LV) epicardial pacing approach

SECONDARY OUTCOMES:
Electrocardiography characteristics - QRS Interval | Procedure Day
  Compare electrocardiography characteristics - QRS Interval measured in seconds between conduction system pacing (CSP) and transthoracic left ventricular (LV) epicardial pacing approach

CONTACTS AND LOCATIONS:
Overall Officials: Naga Venkata K. Pothineni, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

REFERENCES:
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Butter C, Georgi C, Stockburger M. Optimal CRT Implantation-Where and How To Place the Left-Ventricular Lead? Curr Heart Fail Rep. 2021 Oct;18(5):329-344. doi: 10.1007/s11897-021-00528-9. Epub 2021 Sep 8. PMID 34495452
- [Background] Daubert C, Behar N, Martins RP, Mabo P, Leclercq C. Avoiding non-responders to cardiac resynchronization therapy: a practical guide. Eur Heart J. 2017 May 14;38(19):1463-1472. doi: 10.1093/eurheartj/ehw270. PMID 27371720
- [Background] Pothineni NVK, Gondi S, Cherian T, Kovelamudi S, Schaller RD, Lakkireddy D, Gopinathannair R, Deshmukh A. Complications of Cardiac Resynchronization Therapy: Comparison of Safety Outcomes from Real-world Studies and Clinical Trials. J Innov Card Rhythm Manag. 2022 Aug 15;13(8):5121-5125. doi: 10.19102/icrm.2022.130805. eCollection 2022 Aug. PMID 36072440
- [Background] Alonso C, Leclercq C, d'Allonnes FR, Pavin D, Victor F, Mabo P, Daubert JC. Six year experience of transvenous left ventricular lead implantation for permanent biventricular pacing in patients with advanced heart failure: technical aspects. Heart. 2001 Oct;86(4):405-10. doi: 10.1136/heart.86.4.405. PMID 11559679
- [Background] Ahsan SY, Saberwal B, Lambiase PD, Chaubey S, Segal OR, Gopalamurugan AB, McCready J, Rogers DP, Lowe MD, Chow AW. An 8-year single-centre experience of cardiac resynchronisation therapy: procedural success, early and late complications, and left ventricular lead performance. Europace. 2013 May;15(5):711-7. doi: 10.1093/europace/eus401. Epub 2013 Jan 12. PMID 23315159
- [Background] Navia JL, Atik FA, Grimm RA, Garcia M, Vega PR, Myhre U, Starling RC, Wilkoff BL, Martin D, Houghtaling PL, Blackstone EH, Cosgrove DM. Minimally invasive left ventricular epicardial lead placement: surgical techniques for heart failure resynchronization therapy. Ann Thorac Surg. 2005 May;79(5):1536-44; discussion 1536-44. doi: 10.1016/j.athoracsur.2004.10.041. PMID 15854930
- [Background] Sharma PS, Vijayaraman P. Conduction System Pacing for Cardiac Resynchronisation. Arrhythm Electrophysiol Rev. 2021 Apr;10(1):51-58. doi: 10.15420/aer.2020.45. PMID 33936744
- [Background] Chen X, Ye Y, Wang Z, Jin Q, Qiu Z, Wang J, Qin S, Bai J, Wang W, Liang Y, Chen H, Sheng X, Gao F, Zhao X, Fu G, Ellenbogen KA, Su Y, Ge J. Cardiac resynchronization therapy via left bundle branch pacing vs. optimized biventricular pacing with adaptive algorithm in heart failure with left bundle branch block: a prospective, multi-centre, observational study. Europace. 2022 May 3;24(5):807-816. doi: 10.1093/europace/euab249. PMID 34718539
- [Background] Burger H, Pecha S, Hakmi S, Opalka B, Schoenburg M, Ziegelhoeffer T. Five-year follow-up of transvenous and epicardial left ventricular leads: experience with more than 1000 leads. Interact Cardiovasc Thorac Surg. 2020 Jan 1;30(1):74-80. doi: 10.1093/icvts/ivz239. PMID 31633187
- [Background] Kim HR, Lim K, Park SJ, Park JS, Kim JY, Chung S, Jung DS, Park KM, On YK, Kim JS. Thoracoscopic Implantation of Epicardial Left Ventricular Lead for Cardiac Resynchronization Therapy. J Cardiovasc Dev Dis. 2022 May 16;9(5):160. doi: 10.3390/jcdd9050160. PMID 35621871
- [Background] Wu S, Su L, Vijayaraman P, Zheng R, Cai M, Xu L, Shi R, Huang Z, Whinnett ZI, Huang W. Left Bundle Branch Pacing for Cardiac Resynchronization Therapy: Nonrandomized On-Treatment Comparison With His Bundle Pacing and Biventricular Pacing. Can J Cardiol. 2021 Feb;37(2):319-328. doi: 10.1016/j.cjca.2020.04.037. Epub 2020 May 7. PMID 32387225
- [Background] Pujol-Lopez M, Jimenez-Arjona R, Garre P, Guasch E, Borras R, Doltra A, Ferro E, Garcia-Ribas C, Niebla M, Carro E, Puente JL, Vazquez-Calvo S, Invers-Rubio E, Roca-Luque I, Castel MA, Arbelo E, Sitges M, Brugada J, Tolosana JM, Mont L. Conduction System Pacing vs Biventricular Pacing in Heart Failure and Wide QRS Patients: LEVEL-AT Trial. JACC Clin Electrophysiol. 2022 Nov;8(11):1431-1445. doi: 10.1016/j.jacep.2022.08.001. Epub 2022 Oct 26. PMID 36424012
- [Background] Vijayaraman P, Herweg B, Verma A, Sharma PS, Batul SA, Ponnusamy SS, Schaller RD, Cano O, Molina-Lerma M, Curila K, Huybrechts W, Wilson DR, Rademakers LM, Sreekumar P, Upadhyay G, Vernooy K, Subzposh FA, Huang W, Jastrzebski M, Ellenbogen KA. Rescue left bundle branch area pacing in coronary venous lead failure or nonresponse to biventricular pacing: Results from International LBBAP Collaborative Study Group. Heart Rhythm. 2022 Aug;19(8):1272-1280. doi: 10.1016/j.hrthm.2022.04.024. Epub 2022 Apr 30. PMID 35504539
- [Background] Mair H, Sachweh J, Meuris B, Nollert G, Schmoeckel M, Schuetz A, Reichart B, Daebritz S. Surgical epicardial left ventricular lead versus coronary sinus lead placement in biventricular pacing. Eur J Cardiothorac Surg. 2005 Feb;27(2):235-42. doi: 10.1016/j.ejcts.2004.09.029. PMID 15691676